CLINICAL TRIAL: NCT02193516
Title: Identification of Corticomedullary Differentiation Along Different Stage of Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC1413-0250CTIL
Record Dates: First submitted 2014-06-29; First posted 2014-07-17 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Nephropathy
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

SUMMARY:
Corticomedullary differentiation (CMD) abnormality (absent/reversed) is a parameter that can indicate possible nephropathy. The evolution of CMD across gestation had not been well established. Devrendt et al demonstrated the presence of CMD in all fetuses older then 20 weeks. In our study we would like to determine the exact timing of it's sonographic visualisation. This is a prospective study recruiting women between 14-24 week gestation during routine ultrasound screening. A midsagittal image of each kidney will be taken by a single sonographer and examined for the presence of the CMD by two other sonographers blinded to gestational age.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women 14-24 weeks
* singleton pregnancy
* Appropriate for gestational age fetuses
* well dated pregnancy

Exclusion Criteria:

* family history of renal disease
* small /large for gestational age fetuses
* known structural anomalies
* unknown dating

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: pregnant women 14-24 gestational age
Sampling Method: Non-Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
CMD presence | A single exam for each participent. The photos will be reviewed within up to 6 month from examination date

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Hospital, Kfar Saba, Israel